CLINICAL TRIAL: NCT01653301
Title: INTEnsification Radiotherapy With Accelerated Fractionation or ChemoTherapy And Local Excision After 3D External Radio-chemotherapy
Brief Title: Preoperative Downstaging of Extraperitoneal T3 Rectal Cancer: XELOXRT Versus XELACRT. A Multicenter, Phase III Study
Acronym: INTERACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Vincenzo Valentini, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 515(A1144)/2005
Record Dates: First submitted 2012-04-30; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XELOX-RT (Experimental): * Xeloda: 1300 mg/m2 chronomodulated (h 8.00 a.m. 25% of total dose ; h 6.00 p.m. 25% of total dose; h 11.00 p.m. 50% of total dose), during the whole treatment time;
  * Oxaliplatin: 130mg/m2, days 1, 19, 38
  RT: pelvic treatment is the same for both arms: 45 Gy are delivered to the whole pelvis at 1.8 Gy daily, 5 times per week; In the XELOX-RT arm a boost of 5.4 Gy is delivered to the mesorectum corresponding to GTV, at 1.8 Gy daily, in 3 fractions, to a total dose of 50.4 Gy. The boost will be delivered at the end of the irradiation of the pelvis (sequential boost).
  Interventions: Drug: XELOX RT
- XELAC-RT (Active Comparator): Xeloda 1650mg/m2 chronomodulated (h 8.00 a.m. 25% of total dose ; h 6.00 p.m. 25% of total dose; h 11.00 p.m. 50% of total dose) during the whole treatment time.
  RT: pelvic treatment is the same for both arms: 45 Gy are delivered to the whole pelvis at 1.8 Gy daily, 5 times per week.
  In the XEL-ACRT arm a boost of 10 Gy is delivered to the mesorectum corresponding to the GTV, at 1 Gy for fraction to a total dose of 55 Gy, in 10 fractions over 5 weeks, 2 times a week. The daily dose of the boost will be delivered twice a week immediately after the daily dose administered to the pelvis (concomitant boost).
  Interventions: Drug: XELAC RT

INTERVENTIONS:
Drug: XELAC RT — Xeloda 1650mg/m2 chronomodulated (h 8.00 a.m. 25% of total dose ; h 6.00 p.m. 25% of total dose; h 11.00 p.m. 50% of total dose) during the whole treatment time.
  RT: pelvic treatment is the same for both arms: 45 Gy are delivered to the whole pelvis at 1.8 Gy daily, 5 times per week.
  In the XEL-ACRT arm a boost of 10 Gy is delivered to the mesorectum corresponding to the GTV, at 1 Gy for fraction to a total dose of 55 Gy, in 10 fractions over 5 weeks, 2 times a week. The daily dose of the boost will be delivered twice a week immediately after the daily dose administered to the pelvis (concomitant boost).
  Arms: XELAC-RT
Drug: XELOX RT — * Xeloda: 1300 mg/m2 chronomodulated (h 8.00 a.m. 25% of total dose ; h 6.00 p.m. 25% of total dose; h 11.00 p.m. 50% of total dose), during the whole treatment time;
  * Oxaliplatin: 130mg/m2, days 1, 19, 38
  RT: pelvic treatment is the same for both arms: 45 Gy are delivered to the whole pelvis at 1.8 Gy daily, 5 times per week; In the XELOX-RT arm a boost of 5.4 Gy is delivered to the mesorectum corresponding to GTV, at 1.8 Gy daily, in 3 fractions, to a total dose of 50.4 Gy. The boost will be delivered at the end of the irradiation of the pelvis (sequential boost).
  Arms: XELOX-RT

SUMMARY:
* INTERACT study: to evaluate the pathological response rate in cT3 rectal cancer
* LEADER study: to evaluate the impact on local control of local excision

DETAILED DESCRIPTION:
* INTERACT study: to evaluate the pathological response rate evaluated according to TRG scale comparing accelerated radiotherapy on the gross tumour combined plus standard radiotherapy to the pelvis in association with chronomodulated capecitabine (XELACRT arm) versus oxaliplatin added to standard pelvis radiotherapy and same chronomodulated Capecitabine (XELOXRT arm)
* LEADER study: to evaluate the impact on local control of local excision in patients who had a major clinical response evaluated by MRI and confirmed by TRG 1-2 score.

ELIGIBILITY:
INTERACT STUDY

Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma of the rectum.
* Tumour within 12 cm of the anal verge by proctoscopic examination or within 10 cm of the anorectal ring by MRI.
* Clinical stages (UICC 1997): cT2N0-2 low located tumour, cT3 N0-2.
* Resectable disease at the routine examination.
* Age > 18 years.
* Karnofsky Performance Status > 60.
* WBC > 4,000 cells/ml, platelets > 100,000 cells/ml.
* Provision of written informed consent.

Exclusion Criteria:

* Evidence of metastatic (M1) disease. If there were any suspicious findings (i.e. liver metastasis, lung nodule, retroperitoneal adenopathy, etc.) the patient is to be considered as ineligible, unless malignancy is ruled out by tissue documentation (biopsy) before trial therapy is started.
* Previous chemotherapy, immunotherapy, or radiation therapy to the pelvis.
* Multiple primary cancers involving both the colon and rectum that would preclude a patient from being classified as having only rectal cancer.
* Incomplete healing from or other surgery.
* Active inflammatory bowel disease.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
* Cardiovascular disease with a New York Heart Association Functional Status > 2.
* Absolute neutrophil count (ANC) < 4 x 108/L or platelets < 50 x 108/L.
* Measured Creatinine clearance less than 65ml/min. (no drug dose reduction for lower GFR is allowed).
* ALT or AST > 2.5 times the ULRR
* Pregnancy or breastfeeding (women of child-bearing potential).
* Any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
* Any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial.

LEADER STUDY

Inclusion Criteria

* Stage at the diagnosis: cT3N0. T3 patients at the diagnosis with 3 or less enlarged nodes, evaluated by imaging, and without evidence of the same nodes after radiochemotherapy, could be accrued according to Center decision, but will be analyzed separately.
* Patients with cT2N0, low located tumour, otherwise candidates to a Miles surgical procedure, treated by neoadjuvant chemoradiation and with written consensus;
* Major clinical response after chemoradiation, yT0-1N0; yT2N0 could be accrued according to Center decision, but will be analyzed separately.
* Circumferential extension less than 2 quarters;
* Deep ulcer < 2 cm of diameter;
* Provision of written informed consent;
* Biopsies are discouraged for the higher risk of following fistulae in irradiated rectum;

Exclusion Criteria:

* pT3;
* Positive margins;
* TRG 3-5;
* Major adverse features: lymphatic vessel invasion, vascular vessel invasion, perineural invasion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2005-10; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pathological major downstaging | 15-20 weeks after the randomization
  INTERACT study:
  evaluation of T pathological major downstaging, considered as the overall rate of any TRG1 or TRG 2 scored patients;
  LEADER study (optional):
  To evaluate the impact on local control of local excision in patients who had a major clinical response, evaluated by EUS/ MRI, yN0 evaluated by multislice CT / MRI, and confirmed by TRG 1-2 score.

SECONDARY OUTCOMES:
Tumor downstaging | 15-20 weeks after the randomization
  Secondary objectives:
  * Tumour downstaging, evaluated by the comparison of clinical staging before combined modality treatment toward pathological staging.
  * feasibility of a sphincter saving surgical procedure;
  * evaluation of activity of preoperative treatment (clinical response, facultative)
  * post-surgical functional outcome;
  * evaluation of the local control of the disease;
  * estimates (Kaplan-Meier, product limit method) of the disease free survival;
  * Evaluation of adverse events and adverse reactions to treatment, according to both the RTOG and NCI-CTC criteria.
sphincter saving surgery | 15-20 weeks after the randomization
  Secondary objectives:
  * Tumour downstaging, evaluated by the comparison of clinical staging before combined modality treatment toward pathological staging.
  * feasibility of a sphincter saving surgical procedure;
  * evaluation of activity of preoperative treatment (clinical response, facultative)
  * post-surgical functional outcome;
  * evaluation of the local control of the disease;
  * estimates (Kaplan-Meier, product limit method) of the disease free survival;
  * Evaluation of adverse events and adverse reactions to treatment, according to both the RTOG and NCI-CTC criteria.
local control | 15-20 weeks after the randomization
  Secondary objectives:
  * Tumour downstaging, evaluated by the comparison of clinical staging before combined modality treatment toward pathological staging.
  * feasibility of a sphincter saving surgical procedure;
  * evaluation of activity of preoperative treatment (clinical response, facultative)
  * post-surgical functional outcome;
  * evaluation of the local control of the disease;
  * estimates (Kaplan-Meier, product limit method) of the disease free survival;
  * Evaluation of adverse events and adverse reactions to treatment, according to both the RTOG and NCI-CTC criteria.
survival | 15-20 weeks after the randomization
  Secondary objectives:
  * Tumour downstaging, evaluated by the comparison of clinical staging before combined modality treatment toward pathological staging.
  * feasibility of a sphincter saving surgical procedure;
  * evaluation of activity of preoperative treatment (clinical response, facultative)
  * post-surgical functional outcome;
  * evaluation of the local control of the disease;
  * estimates (Kaplan-Meier, product limit method) of the disease free survival;
  * Evaluation of adverse events and adverse reactions to treatment, according to both the RTOG and NCI-CTC criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy, Italy

REFERENCES:
- [Derived] Valentini V, Gambacorta MA, Cellini F, Aristei C, Coco C, Barbaro B, Alfieri S, D'Ugo D, Persiani R, Deodato F, Crucitti A, Lupattelli M, Mantello G, Navarria F, Belluco C, Buonadonna A, Boso C, Lonardi S, Caravatta L, Barba MC, Vecchio FM, Maranzano E, Genovesi D, Doglietto GB, Morganti AG, La Torre G, Pucciarelli S, De Paoli A. The INTERACT Trial: Long-term results of a randomised trial on preoperative capecitabine-based radiochemotherapy intensified by concomitant boost or oxaliplatin, for cT2 (distal)-cT3 rectal cancer. Radiother Oncol. 2019 May;134:110-118. doi: 10.1016/j.radonc.2018.11.023. Epub 2019 Feb 7. PMID 31005204